CLINICAL TRIAL: NCT02441907
Title: Predictors of Treatment Response to Aflibercept and Aqueous Cytokine Levels in Treatment Naïve Patients With Diabetic Macular Edema
Brief Title: Predictors of Treatment Response to Aflibercept and Aqueous Cytokine Levels in Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aflibercept Cytokine DME
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Ocular Cytokines; Triamcinolone Acetonide
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aflibercept treatment (Other): aflibercept, 40 mg/mL Solution for Intravitreal Injection
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept
  Other Names: Eylea

SUMMARY:
Diabetic macular edema refers to swelling (fluid accumulation) in the center of the retina. The retina is like the film of a camera and is located in the back of the eye. This condition can develop in diabetics where swelling results from leaking of fluid from the blood vessels of the eye, into the center of the retina, the macula. If left untreated, this can affect central vision. The current standard treatment for diabetic macular edema includes medications injected directly into the eye (intravitreal injections) and laser eye treatment. The drugs that are injected directly into the eye are known as anti-Vascular Endothelial Growth Factor (anti-VEGF) agents which help to reduce the leaking. However, response in patients to these anti-VEGF drugs can vary and examination of predictive factors is required. This particular study examines cellular factors called cytokines in patients receiving aflibercept, a type of anti-VEGF drug, in the hopes of detecting changes in cytokines that can predict treatment response amongst groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above
* Presence of Non Proliferative Diabetic Retinopathy (NPDR)
* Treatment Naïve patients with DME with central macular thickness of 310μm or more on SD-OCT (cirrus)
* Subjects with Type I or II diabetes mellitis
* Willing and able to provide informed consent for participation in the study

Exclusion Criteria:

* Proliferative diabetic retinopathy in the study eye or PRP within the last 12 months or anticipated PRP in the next 6 months
* Uncontrolled glaucoma
* History of intraocular surgery within 3 months in the study eye
* History of vitrectomy surgery
* Laser treatment within 3 months of study eye
* Vitreomacular traction, epiretinal membrane or any other maculopathy in the study eye
* Prior intravitreal injection within the past 6 months
* Known allergy to the study drug or fluorescein
* History of stroke or AMI within 6 months of enrollment
* Patients receiving dialysis for renal failure
* Patients currently on systemic immunosuppression
* Patients on two or more class of medication for glaucoma in study eye
* Patients with tuberculosis
* Patients who are pregnant.
* Unwilling or unable to follow or comply with all study related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in cytokine levels (picograms per mL) between baseline aflibercept injection and at 1, 2, and 3 months | 3 months

SECONDARY OUTCOMES:
Relation of baseline aqueous cytokine levels to baseline Snellen BCVA in response to aflibercept | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev Muni, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital Eye Clinic, Toronto, Ontario, Canada